CLINICAL TRIAL: NCT02354183
Title: Commitment and Motivation in a Brief DBT Intervention for Self Harm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Michelle Leybman, Clinical Psychologist, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 070/2013
Record Dates: First submitted 2014-12-10; First posted 2015-02-03 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2017-02

CONDITIONS: Psychological Orientation; Acceptance Processes
Keywords: Commitment strategies; Motivation; DBT skills; Self-harm; Brief intervention
MeSH Terms: conditions — Orientation, Spatial; Behavior; Self-Injurious Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Commitment (Experimental): A 1-hour orientation session consisting of DBT commitment strategies plus psychoeducation. Therapists will also use commitment strategies to discuss goals related to self-harm. The psychoeducation will consist of information about DBT's biosocial theory and about why people self-harm. All participants will complete a DBT skills training group after their orientation.
  Interventions: Behavioral: DBT Skills Training
- Psychoeducation (Active Comparator): A 1-hour orientation session consisting of psychoeducation only. The psychoeducation will consist of information about DBT's biosocial theory and about why people self-harm. All participants will complete a DBT skills training group after their orientation.
  Interventions: Behavioral: DBT Skills Training

INTERVENTIONS:
Behavioral: DBT Skills Training — Based on Linehan's (1993) manualized DBT approach, the brief DBT skills training group covers will cover five skills: wise mind, TIP skills, distraction, mindfulness of the current emotion, and opposite to emotion action.

SUMMARY:
Research suggests that individuals with Borderline Personality Disorder (BPD) experience low motivation for change (Skodal, Buckley, & Charles, 1983). Dialectical Behavior Therapy (DBT; Linehan, 1993) includes commitment strategies that are designed to improve motivation. No studies have examined the effectiveness of these strategies. The proposed study will evaluate the efficacy of a brief DBT intervention consisting of commitment strategies plus skills training for people who self-harm. Participants will be randomly assigned to either a single orientation session of (1) commitment strategies plus psychoeducation or (2) psychoeducation. Immediately following their orientation session, all participants will be enrolled in a 90 minute group skills training session. Primary outcomes include autonomous motivation and frequency of self harm behaviours. Assessments will be conducted at six time points: baseline, after the initial orientation session, after the skills training group session, and at one week, one month, and three month follow-up

DETAILED DESCRIPTION:
Client motivation is related to therapeutic change (Ryan, Lynch, Vansteenkiste, & Deci) and low motivation is a pervasive issue for clients with BPD (e.g., Skodal et al., 1983). DBT (Linehan, 1993) is an effective treatment for BPD and was developed in part to address client motivation. Within DBT there are commitment strategies that are used to help clients establish clear goals and increase motivation to work on them. These strategies were designed to help people commit to eliminating self-harm as well as other behaviours. People are more motivated to work effectively towards goals for which they are autonomously motivated (Deci & Ryan, 2000). Despite their importance in DBT, commitment strategies have never been studied. This study will examine whether commitment strategies are associated with an increase in autonomous motivation and a decrease in self harm behaviour.

This research will address two primary questions: 1) Are commitment strategies associated with an increase in autonomous motivation to decrease self-harm behaviour?; and 2) Does autonomous motivation mediate a relationship between commitment strategies and change in self-harm behaviour? The investigators will also address a secondary question related to predictors of autonomous motivation. Our hypotheses are as follows: 1) The group receiving psychoeducation enhanced with commitment strategies will have higher levels of autonomous motivation compared to the psychoeducation control group; and 2) autonomous motivation will mediate the relationship between commitment strategies and decreases in self harm behaviour. Additionally, autonomy support, low therapist judgment, and goal concordance between client and therapist will independently contribute to predicting client autonomous motivation.

Research in this area is needed in light of the challenges presented by the low motivation that often characterizes individuals with borderline traits who engage in self-harm behaviour. No studies to date have examined DBT's commitment strategies, thus, the effect of these treatment strategies is unknown and needs to be established. Additionally, identifying specific variables that are associated with motivation to eliminate self-harm will help inform the refinement treatment strategies. Finally, few studies have examined the role of autonomous motivation and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Has a valid health card issued by a Canadian province or Canadian student organization (ie: UHIP)
2. Has had at least 3 self-harm episodes (either suicidal or non-suicidal) in the past 5 years, including at least 1 in the past eight weeks
3. Is literate in English
4. Absence of 4 or more formal weeks of DBT in the past year (individual or group therapy components)
5. Indicates absence of knowledge of the DBT Skills
6. Is able to attend all sessions on scheduled study day

Exclusion Criteria:

1) Evidence of organic brain syndrome or mental retardation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2015-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change in Autonomous and Controlled Motivation | From baseline until 3 months following the completion of the 1-day intervention (i.e., average of 3 months)
  Autonomous and controlled motivation will be assessed using the Autonomous and Controlled Motivation for Treatment Questionnaire (Zuroff et al., 2005).

SECONDARY OUTCOMES:
Change in Frequency and severity of self-harm behaviour | From baseline until 3 months following the completion of the 1-day intervention (i.e., average of 3 months)
  The frequency and severity of self-harm behaviour will be assessed using the Deliberate Self-Harm Inventory, a 17-item self-report questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Leybman, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617
- See also: Information about research at the Centre for Addiction and Mental Health, Canada's largest mental health and addiction teaching hospital, fully affiliated with the University of Toronto, and a PAHO/WHO Collaborating Centre — http://www.camh.ca/en/research